CLINICAL TRIAL: NCT06492122
Title: A Phase 1, First-in-Human, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of [225Ac]Ac-FL-020 in Participants With mCRPC.
Brief Title: Study With [225Ac]Ac-FL-020 in mCRPC Participants
Acronym: ProTACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Full-Life Technologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-020-001
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Safety; RP2D; Pharmacokinetics; Dosimetry; Preliminary efficacy; Dose escalation; Dose expansion; PSMA; mCRPC; Prostate; Radiopharmaceutical; RDC; Phase I; Actinium-225; Full-Life; RLT; ProTACT
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [225Ac]Ac-FL-020 (Experimental): Treatment with [225Ac]Ac-FL-020 administered intravenously. 10 patients will also receive [111In]In-FL-020 for dosimetry purposes.
  Interventions: Drug: [225Ac]Ac-FL-020; Drug: Blood samples for PK; Drug: [111In]In-FL-020; Procedure: Blood and urine samples collection; Procedure: SPECT/CT images

INTERVENTIONS:
Drug: [225Ac]Ac-FL-020 — [225Ac]Ac-FL-020 injected intravenously
Drug: Blood samples for PK — Following the first injection of [225Ac]Ac-FL-020, blood samples after treatment will be collected for PK evaluation.
Drug: [111In]In-FL-020 — A dose of [111In]In-FL-020 will be injected prior to the first dose of [225Ac]Ac-FL-020 for dosimetry evaluation
Procedure: Blood and urine samples collection — For dosimetry evaluation and urine excretion assessment, blood and urine samples will be collected after the injection of [111In]In-FL-020
Procedure: SPECT/CT images — For dosimetry evaluation, SPECT/CTs will be performed following the injection of [111In]In-FL-020.

SUMMARY:
The purpose of this study is to evaluate the safety, therapeutic effect, and pharmacokinetics of [225Ac]Ac-FL-020 in participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The aim of this Phase 1, First-in-Human, Open-label Trial is to evaluate the safety, tolerability, pharmacokinetics, and efficacy of [225Ac]Ac-FL-020 as a single agent in participants with metastatic Castration-Resistant Prostate Cancer (mCRPC). [111In]In-FL-020 serves as a surrogate for 225Ac-FL-020 for dosimetry purposes. The trial is divided into two parts: dose escalation in Part 1 and cohort expansion in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic CRPC.
2. Age ≥ 18 years.
3. Signed informed consent, and able and willing to comply with protocol requirements prior to any study procedures.
4. Patients must have a life expectancy >3 months.
5. All patients are required to have one or more positive lesions detected by PSMA-PET/CT scan
6. Documented progression of the disease based on the Investigator judgement
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Have a castrate serum testosterone < 50 ng/dL or <1.7 nmol/L. Patients must continue primary androgen deprivation with an LHRH analogue (agonist/antagonist) if they have not undergone bilateral orchiectomy.
9. Have previously been treated with at least one of the following:

   1. Androgen receptor signaling inhibitor (such as enzalutamide).
   2. CYP 17 inhibitor (such as abiraterone acetate).
10. Patients must have been previously treated with at least 1, but no more than 2 previous taxane regimens. Note: In cases where patients are unwilling to undergo taxane therapy due to concerns regarding its potential toxicity, enrollment of patients previously not treated with taxane might be considered after careful evaluation by the investigator. In such cases, patients will be fully informed about the potential benefits of taxane therapy, including its role in prolonging survival.
11. Adequate organ function as defined by:

    1. Absolute neutrophil count (ANC) ≥2 x 10^9/L (2000/µL),
    2. Hemoglobin ≥9.0 g/dL,
    3. Platelets ≥90 x 10^9/L (90 000/µL),
    4. Serum albumin >3g/dL
    5. Aspartate aminotransferase (AST) ≤2.5 x ULN; alanine aminotransferase (ALT) ≤2.5 x ULN (AST, ALT ≤5 x ULN if liver metastases are present),
    6. Serum total bilirubin ≤1.5 x ULN (≤5 x ULN if liver metastases present)
    7. Creatinine clearance ≥60 mL/min calculated using a standard Cockcroft and Gault formula.
    8. Q wave to T wave (QT) interval corrected for heart rate (QTc) <470 ms

Exclusion Criteria:

1. Patients with known brain metastases.
2. Grade 3 Cystitis infective and non-infective.
3. Severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the study treatment administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for enrollment in this study.
4. More than 1 prior treatment with PSMA-targeted radioconjugate.
5. Previous treatment with Actinium-225, Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, or hemi-body irradiation or any other radionuclide therapy except [177Lu]Lu-PSMA-617 and Radium-223.
6. Radium-223 within 6 months prior to the first study treatment administration.
7. Prior radioconjugate treatment within 6 weeks prior to first study treatment administration. Adverse events from prior radioconjugate treatment must be resolved or reduced to grade 1 prior to the first study treatment administration.
8. More than 6 administrations of previous radioconjugate treatment.
9. Any systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 6 weeks prior to the first study treatment administration. Patients on a stable bisphosphonate or denosumab regimen for 30 days prior to first study treatment administration are eligible.
10. Evidence of superscan in the baseline bone scan.
11. Any investigational agents within 6 weeks prior to the first study treatment administration.
12. Radiotherapy: external beam radiotherapy that encompasses >30% of bone marrow completed less than 6 weeks or focal radiation completed less than 2 weeks, prior to the first study treatment administration.
13. Major surgery (not including placement of vascular access device or tumor biopsies) within 6 weeks prior to first dose of the study treatment, or no recovery from side effects of such intervention.
14. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
15. Known hypersensitivity to the components of the study therapy or its analogs.
16. Enrollment in another interventional clinical study.
17. Any persistent xerostomia or dry eyes from previous treatment
18. Persistent prior AEs > Grade 1 from prior anti-cancer therapies.
19. Significant cardiac disease, such as recent (within six months prior to first dose of the study treatment) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension, uncontrolled cardiac arrhythmias, severe aortic stenosis.
20. History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within 6 months prior to first dose of the study treatment.
21. Known active infection requiring therapy, including known active infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or SARS-CoV-2
22. Prior history of malignancy other than inclusion diagnosis within three years prior to first dose of the study treatment
23. Known history of myelodysplastic syndrome.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are male with mCRPC
Enrollment: 50 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose escalation: Incidence of Dose-Limiting Toxicities (DLTs). | 28 days after the first injection of [225Ac]Ac-FL-020
  RP2D
Dose escalation and dose expansion: Type, frequency and severity of adverse events (AEs) and serious adverse events (SAEs) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | From ICF signature and up to 42 days after the last dose of study treatment for all AE and SAE. Then only the AE/SAE suspected to be related to the study treatment will be reported.

SECONDARY OUTCOMES:
Dose escalation and dose expansion: Absorbed doses | During one week following the injection of [111In]In-FL-020
  Absorbed doses in different organs and tumors
Peak Plasma Concentration (Cmax) | During one week following the first injection of [225Ac]Ac-FL-020
  Pharmacokinetics
Area Under the Plasma concentration versus time curve | During one week following the first injection of [225Ac]Ac-FL-020
  Pharmacokinetics
Overall response rate | 2 years
  Anti-tumor activity via imaging assessments and PSA levels
Disease Control Rate | 2 years
  Anti-tumor activity via imaging assessments and PSA levels
Best Overall response | 2 years
  Anti-tumor activity via imaging assessments and PSA levels
Progression Free Survival | 2 years
  Anti-tumor activity via imaging assessments and PSA levels
Overall Survival | 2 years
  Anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Full-Life Technologies GmbH, Study Director — Full-Life Technologies GmbH
Locations (9):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Chao Family Comprehensive Cancer Center, Irvine, California
  - University of Stanford, Stanford, California
  - University of Virginia Cancer Center, Charlottesville, Virginia
- Australia (3):
  - Princess Alexandra Hospital, Brisbane
  - Genesiscare Murdoch, Murdoch
  - MacQuarie University Clinical Trial Unit, Sydney
- Beijing Cancer Hospital, Beijing, China
- Ankara Üniversitesi Tıp Fakültesi Cebeci Hastanesi Nükleer Tıp Anabilim Dalı, Ankara, Turkey (Türkiye)